CLINICAL TRIAL: NCT02700295
Title: Long Term Effects of Multifocal Orthokeratology on Corneal and Choroidal Structures in Healthy Subjects With Myopia- A Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, MD, PhD, Medical University of Vienna
Other Study IDs: OPHT-260514
Record Dates: First submitted 2016-02-24; First posted 2016-03-07 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Myopia
Keywords: Orthokeratology
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Orthokeratology contact lens group
  Interventions: Device: Orthokeratology lens

INTERVENTIONS:
Device: Orthokeratology lens

SUMMARY:
Orthokeratology has the benefit for slowing down myopia progression and enabling unaided vision during the day. To investigate proposed possible changes of conventional and multifocal orthokeratology in the cornea and choroid this study will image both structures with high resolution optical coherence tomographs over a six month period. Findings will help to plan larger trials over a longer period of time in adults and teenagers.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged over 18 years
* Myopia defined as between -1D and -6 D with an increase of 0.5D within the last 18months prior to inclusion
* Prospect orthokeratology contact lens wearers
* Normal findings in the slit lamp examination, no corneal pathologies

Exclusion Criteria:

* Participation in a clinical trial in the previous 3 weeks
* Presence of any abnormalities (such as refractive surgery) preventing reliable measurements as judged by the investigator
* Current contact lens wearers
* Pregnancy, planned pregnancy or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy volunteers
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2016-02; Primary Completion 2023-09 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Quantitative changes in the corneal thickness | 1 year
Qualitative changes in the corneal structure | 1 year

SECONDARY OUTCOMES:
Quantitative changes in the choroidal thickness | 1 year
Qualitative changes in the choroidal structure | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Medical Physics and Biomedical Engineering, Medical University of Vienna, Vienna, Austria